CLINICAL TRIAL: NCT04451148
Title: Gut Microbiome As Target of Intervention Against Obesity and Metabolic Syndrome
Brief Title: Gut Microbiome and Obesity
Acronym: MATOMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, Associate Professor, Federico II University
Other Study IDs: 103/20
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Obesity, Childhood; Metabolic Syndrome
MeSH Terms: conditions — Pediatric Obesity; Metabolic Syndrome | interventions — Adiposity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese subjects: Subjects with obesity
  Interventions: Other: Obese with or without metabolic syndromesubjects
- Obese plus metabolic syndrome subjects: Subjects with obesity and metabolic syndrome
  Interventions: Other: Obese with or without metabolic syndromesubjects
- Healthy controls: Otherwise healthy subjects

INTERVENTIONS:
Other: Obese with or without metabolic syndromesubjects — Children with obesity and with or without metabolic syndrome
  Groups: Obese plus metabolic syndrome subjects; Obese subjects

SUMMARY:
Pediatric obesity is a risk factor for the onset of obesity in adulthood and is a risk factor for various chronic non-communicable diseases. Metabolic syndrome (MS) is the name for a group of risk factors that increase cardiovascular risk and other health problems characterized by the presence of abdominal obesity, dyslipidemia, hyperglycaemia and high blood pressure. Numerous preclinical and clinical data suggest a potential role of the intestinal microbiota in these diseaes. Unfortunately, comparative studies of the gut microbiota are still scarce in pediatric subjects suffering from obesity than obesity complicated by MS. The aim is to study the metagenomics and metabolomics characteristics of the intestinal microbiota in obese children/adolescents with or without MS, that could provide useful data for innovative intervention strategies for these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 10-16 years,
* diagnosis of obesity or obesity complicated by metabolic syndrome
* healthy controls

Exclusion Criteria:

* Age at enrollment < 10 or >16 years,
* concomitant presence of chronic diseases,
* neoplasms,
* immunodeficiencies,
* chronic infections,
* autoimmune diseases,
* chronic inflammatory bowel diseases,
* celiac disease, -genetic-metabolic diseases, -
* cystic fibrosis
* chronic lung diseases,
* malformations of the cardiovascular/respiratory/gastrointestinal system,
* neuropsychiatric disorders
* neurological pathologies,
* assumption of antibiotics and/or pre/pro/synbiotics
* onset of diarrhea or acute gastrointestinal disease during the 12 weeks prior to enrollment.

Ages: 10 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Children/adolescents of both sexes, aged between 10-16 years, with obesity, obesity complicated by metabolic syndrome and healthy controls observed at Pediatrics Section of Department of Translational Medical Sciences (University of Naples Federico II)
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of metagenomic characteristics of the intestinal microbiota in subjects with obesity, obesity complicated by metabolic syndrome and healthy controls | at enrollment
  Evaluation of gut microbiota composition

SECONDARY OUTCOMES:
Concentration of metabolomic characteristics of the intestinal microbiota in subjects with obesity, obesity complicated by metabolic syndrome and healthy controls | at enrollment
  Evaluation of butyrate
Concentration of the metabolomic characteristics of the intestinal microbiota in subjects with obesity, obesity complicated by metabolic syndrome and healthy controls | at enrollment
  Evaluation of acetate
Concentration of the metabolomic characteristics of the intestinal microbiota in subjects with obesity, obesity complicated by metabolic syndrome and healthy controls | at enrollment
  Evaluation of propionate
Concentration of the metabolomic characteristics of the intestinal microbiota in subjects with obesity, obesity complicated by metabolic syndrome and healthy controls | at enrollment
  Evaluation of indole

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided